CLINICAL TRIAL: NCT05204771
Title: Prenatal Ultrasound Assessment of the Relative Position of the Superior Mesenteric Artery and Vein to Define the Status of Digestive Rotation: a Prenatal Tool of Intestinal Malrotation Diagnosis?
Brief Title: Prenatal US Assessment of Superior Mesenteric Vessels for Digestive Rotation
Acronym: SMA
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0683
Record Dates: First submitted 2021-11-24; First posted 2022-01-24 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Singleton-Merten Syndrome; Postnatal Complication
Keywords: Evolution and complication; Mesenteric vessels positionning; 3rd ultrasound examination; Pediatric follow up +/- treatment
MeSH Terms: conditions — Singleton Merten syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Normal foetus: All pregnant women reffered for 3rd trimester routine ultrasound examination without any fetal abnormality
  Interventions: Other: Ultrasound exam; Other: Postnatal abdominal ultrasound; Other: Pediatric Follow up

INTERVENTIONS:
Other: Ultrasound exam — Ultrasound exam
Other: Postnatal abdominal ultrasound — Postnatal abdominal ultrasound
Other: Pediatric Follow up — Pediatric Follow up

SUMMARY:
Digestive malrotation is an anatomical anomaly of the positionning of the mesenteric vessels and the digestive tract that can lead in some form to a dangerous neonatal complication: intestinal volvulus. This requires emergency surgery with a risk of digestive resection. Visualizing during pregnancy the normal or abnormal anatomical positionning of the mesenteric vessels could make it possible to diagnose this malrotation and prevent the occurrence of this complication.

The aim of the study is ti evaluate the ability to identiy prenataly during ultrasound examination, the relative positionning of the fetal mesenteric vessels, and then to correlate it with the real postnatal positionning (gold standard)

DETAILED DESCRIPTION:
* Prenatal US assessment of mesenteric vessels positioning (relative position of the vein vs artery) during routine 3rd trimester US scan
* Description of various anatomical situation
* Comparison of this prenatal positioning with postnatal positioning obtained through abdominal ultrasound examination. Post-natal ultrasound being the gold standard

ELIGIBILITY:
Inclusion criteria:

* Pregnant women attending for 3rd trimester ukltrasound
* Uneventfull pregnancy
* No foetal malformation
* Singleton pregnancy
* Age >18 years

Exclusion criteria:

- Other condition

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant women attending for 3rd timester scan
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Prenatal ultrasound evaluation | day 1
  Prenatal ultrasound evaluation, during 3rd trimester routine scan, of the relative positioning of the superior mesenteric vein in comparison to the superior mesenteric artery

SECONDARY OUTCOMES:
Prenatal ultrasound evaluation | day 1
  Prenatal ultrasound evaluation, during 3rd trimester routine scan, of the relative positioning of the superior mesenteric artery in comparison to the superior mesenteric vein
Prenatal ultrasound evaluation | day 1
  Prenatal ultrasound evaluation, during 3rd trimester routine scan, of the relative positioning of the superior mesenteric artery in comparison to the superior mesenteric aorta

CONTACTS AND LOCATIONS:
Overall Officials: Florent FUCHS, PhD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC